CLINICAL TRIAL: NCT05915962
Title: Biological Characterization Study of an Autograft Nanofat (Nanocarabio)
Acronym: Nanocarabio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-A01605-34
Record Dates: First submitted 2023-06-12; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Rhizarthrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteer for an autograft (Experimental): Collecting and preparing a Nanofat-type autograft using a special kit.
  Interventions: Procedure: collecting a Nanofat-type microfat autograft

INTERVENTIONS:
Procedure: collecting a Nanofat-type microfat autograft — Collecting and preparing a Nanofat autograft.
  The protocol provides for the fat sample to be taken in a doctor's office during a consultation. The preparation will then be carried out at the MEARY center for cell and gene therapy of the AP-HP, at the Saint Louis hospital in Paris.

SUMMARY:
Rhizarthrosis (trapeziometacarpal osteoarthritis) is the most common primary osteoarthritis of the hand, and a source of major functional impact, as it affects the thumb. Non-surgical therapeutic means are currently limited to wearing an immobilization splint, analgesics and oral non-steroidal anti-inflammatory drugs. These symptomatic treatments are of limited effectiveness and do not prevent from progression of the osteoarthritis disease. The most effective treatments currently recognized are surgical, but they also have their limits.

Cell therapy is considered as a promising approach to treat tissue damage including osteoarthritis. Mesenchymal stromal cells are excellent candidates for achieving this type of result, because they can differentiate into the different tissues from the mesoderm (cartilage, bone, muscle, tendons, fat, dermis, conjunctive matrix, etc.). In addition, unlike cells from the embryonic cord, the risk of teratoma or tumor does not exist.

Mesenchymal stem cells have regenerative and immunomodulatory properties but the methods of collection, preparation, combination with substances such as hyaluronic acid, or PRP, or platelet concentrates, will obviously influence the effectiveness of the results. .

Nanofat autografts are obtained in a simple way, in a closed circuit, preserving the stromal mesenchymal cells in large numbers with a minimum impact on the cellular elements. The preparation remains simple and inexpensive, but it is nevertheless necessary to characterize these emulsified preparations biologically before using them as cell therapy.

The main objective of this study is to characterize a nanofat autograft on a biological level.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers, men or women, aged at least 20 to 75 years old.
2. BMI ≥ 20 Kg/m² (in order to have adipose tissue in quantity sufficient)
3. Volunteers who signed an informed consent
4. Hemoglobinemia > 10g/dl
5. Negative Beta-HCG assay
6. Volunteers benefiting from or affiliated to a social security scheme

Exclusion Criteria:

1. Thrombocytopenia < 150 G/L
2. Thrombocytosis > 450 G/L
3. Known thrombopathy
4. TP < 70%
5. APT Patient/Control ratio > 1.20
6. Anemia < 10g/dl
7. Taking antiplatelet, aspirin, anti vitamin K dating less than 15 days before inclusion
8. Fever or recent infection (bacterial or viral) dating from less than a month
9. Autoimmune diseases confirmed by questioning, or clinical and/or biological elements (inflammatory assessment: VS, CRP, fibrinogen) and may interfere with the quality of autograft
10. Inflammatory arthritis
11. Microcrystalline Arthritis
12. Immunodeficiency
13. Current or chronic infectious diseases (viral or bacterial) attested by clinical elements and/or biological (inflammatory assessment: ESR, CRP, Fibrinogen)
14. Malignant tumor under treatment or history of malignant tumor
15. BMI < 20 Kg/m²
16. Contraindication to local anesthesia or surgery
17. Pregnant or breastfeeding women
18. Adults protected by law (under guardianship and guardianship)
19. People participating simultaneously in another research involving the human person
20. Miners
21. Persons staying in a health or social establishment
22. People in an emergency situation
23. Persons deprived of liberty
24. Persons not covered by a social security scheme

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Appearance of nanofat autografts | one month
  Expected specification: colorless to slightly yellow
Flow cytometry count of the following cells : leukocytes, stromal celles and endothelial cells | one month
  * Leukocytes (CD45+): 15 to 55%
  * Stromal cells (CD45-CD34bright CD146-CD90+): 40 to 60%
  * Endothelial cells (CD34bright CD146+CD45-): 1 to 19%
Functionality of nanofat autografts | one month
  Expected specification: CFU-F > 10 per 1000 nucleated cells
Microbiological sterility of nanofat autografts | one month
  expected specification: negative

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Paul d'Egine, Champigny-sur-Marne, France